CLINICAL TRIAL: NCT05630833
Title: A Phase III, Multicenter, Randomized, Active Reference, Double Blind, Double-dummy Study in Japanese Female Participants to Evaluate the Efficacy and Safety of Gepotidacin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)
Brief Title: A Study to Investigate the Efficacy and Safety With Gepotidacin in Japanese Female Participants With Uncomplicated Urinary Tract Infection (Acute Cystitis)
Acronym: EAGLE-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214144
Record Dates: First submitted 2022-11-23; First posted 2022-11-30 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Urinary Tract Infections
Keywords: Acute cystitis; Efficacy; Gepotidacin; Nitrofurantoin; Urinary Tract Infection; Japanese Female
MeSH Terms: conditions — Urinary Tract Infections | interventions — gepotidacin; Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gepotidacin + Placebo (Experimental)
  Interventions: Drug: Gepotidacin; Drug: Placebo
- Nitrofurantoin + Placebo (Active Comparator)
  Interventions: Drug: Nitrofurantoin; Drug: Placebo

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be administered.
  Arms: Gepotidacin + Placebo
Drug: Nitrofurantoin — Nitrofurantoin will be administered.
  Arms: Nitrofurantoin + Placebo
Drug: Placebo — Placebo will be administered.

SUMMARY:
The purpose of this study is to evaluate the consistency of therapeutic response of gepotidacin in female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at baseline that all are susceptible to nitrofurantoin in Japan, with that from global studies (Studies 204989 [NCT04020341] and 212390 [NCT04187144]).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body weight >=40 kilograms (kg).
* The participant has 2 or more of the following clinical signs and symptoms of acute cystitis with onset less than (<) 96 hours prior to study entry: dysuria, frequency, urgency, or lower abdominal pain.
* The participant has nitrite or pyuria (greater than [>]15 white blood cell [WBC]/high-power field [HPF] or the presence of 3 plus (+) /large leukocyte esterase) from a pretreatment clean-catch midstream urine sample based on local laboratory procedures.
* The participant is capable of giving signed informed consent/assent.

Exclusion Criteria:

* The participant resides in a nursing home or dependent care type facility.
* The participant has a body mass index >=40.0 kilogram per meter square (kg/m^2) or a body mass index >=35.0 kg/m^2 and is experiencing obesity-related health conditions such as uncontrolled high blood pressure or uncontrolled diabetes.
* The participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of treatment failure and/or complications.
* The participant has any of the following:

  * Poorly controlled asthma or chronic obstructive pulmonary disease; Acute severe pain; Active peptic ulcer disease; Parkinson disease; Myasthenia gravis; a history of seizure disorder requiring medications for control (this does not include a history of childhood febrile seizures); Or
  * Known acute porphyria.
  * Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention.
* The participant has a known glucose-6-phosphate dehydrogenase deficiency.
* The participant, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* The participant has acute uncomplicated cystitis that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to Pseudomonas aeruginosa or Enterobacterales (other than E. coli) as the contributing pathogen.
* The participant has symptoms known or suspected to be caused by another disease process, such as asymptomatic bacteriuria, overactive bladder, chronic incontinence, or chronic interstitial cystitis, that may interfere with the clinical efficacy assessments or preclude complete resolution of acute cystitis symptoms.
* The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease (e.g., polycystic renal disease), or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract (e.g., chronic vesicoureteral reflux, detrusor insufficiency).
* The participant has an indwelling catheter, nephrostomy, ureter stent, or other foreign material in the urinary tract.
* The participant who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptom onset >=96 hours before study entry, or a temperature >=38 Degrees Celsius [°C], flank pain, chills, or any other manifestations suggestive of upper UTI.
* The participant has known anuria, oliguria, or significant impairment of renal function (creatinine clearance <60 milliliters per minute (mL/min) or clinically significant elevated serum creatinine as determined by the investigator).
* The participant presents with vaginal discharge at Baseline (e.g., suspected sexually transmitted disease).
* The participant has congenital long QT syndrome or known prolongation of the corrected QT (QTc) interval.
* The participant has uncompensated heart failure.
* The participant has severe left ventricular hypertrophy.
* The participant has a family history of QT prolongation or sudden death.
* The participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or brady arrhythmia within the last 12 months.
* The participant is taking QT-prolonging drugs or drugs known to increase the risk of torsades de pointes (TdP) per the www.crediblemeds.org. "Known Risk of TdP" category at the time of her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor.
* For any participant >=12 to <18 years of age, the participant has an abnormal ECG reading at Baseline.
* The participant has a QTc >450 msec or a QTc >480 msec for participants with bundle branch block.
* The participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.
* The participant has a known alanine aminotransferase (ALT) value >2 times upper limit of normal (ULN).
* The participant has a known total bilirubin value >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* The participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice.
* The participant has a previous history of cholestatic jaundice/hepatic dysfunction associated with nitrofurantoin.
* The participant has received treatment with other systemic antimicrobials or systemic antifungals within 1 week before study entry.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 380 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Japan (13):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 380 participants were enrolled in the study. Of these, 374 participants were included in the Intent-to-treat (ITT) population. The ITT population excluded 6 participants from a site with Good Clinical Practice (GCP) violation and therefore not a part of analysis population.
Groups:
- Gepotidacin: Participants with uncomplicated urinary tract infection (uUTI) (acute cystitis) randomized to receive gepotidacin 1500 milligram (mg) (2*750 mg, tablets), twice daily (BID), orally on Day 1 to Day 5. The total daily dose of gepotidacin received was 3000 mg. Participants also received 1 capsule of placebo matched with nitrofurantoin BID, orally on Day 1 to Day 5. All doses were administered after food consumption and with water.
- Nitrofurantoin: Participants with uncomplicated urinary tract infection (acute cystitis) randomized to receive nitrofurantoin 100 mg capsule, BID, orally on Day 1 to Day 5. The total daily dose of nitrofurantoin received was 200 mg. Participants also received 2 tablets of placebo matched with gepotidacin BID, orally on Day 1 to Day 5. All doses were administered after food consumption and with water.
Period: Overall Study
Arm/Group | Gepotidacin | Nitrofurantoin
Started (Enrolled) | 286 | 94
ITT Population (All participants (except for 6 participants from the site with GCP violation) were randomly assigned to the study treatment.) | 281 | 93
Microbiological ITT (Micro-ITT) (All participants (except for 6 participants from the site with GCP violation) were randomly assigned to study treatment who received at least 1 dose of study treatment and had a qualifying baseline uropathogens (UP), from a quantitative bacteriological culture of a pretreatment clean-catch midstream urine specimen.) | 88 | 29
Micro-ITT NTF-S (Participants in micro-ITT population whose baseline qualifying bacterial UP were susceptible to nitrofurantoin (NTF-S).) | 83 | 25
Micro-ITT MDR (Microbiological intent-to-treat multi drug resistant (Micro-ITT MDR) population included all participants in the micro-ITT Population who had any qualifying baseline bacterial UP that were resistant to two or more classes of antimicrobials.) | 18 | 3
Safety (Safety Population included all randomized participants (except for 6 participants from the site with GCP violation) who received at least 1 dose of study treatment.) | 281 | 93
Completed | 279 | 92
Not Completed | 7 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: ITT population: All participants (except for 6 participants from the site with GCP violation) were randomly assigned to the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gepotidacin | Nitrofurantoin | Total
Number analyzed (Participants) | 281 | 93 | 374
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 44.9 (18.78) | 46.4 (19.21) | 45.2 (18.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 93 | 374
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 281 | 93 | 374
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Therapeutic Response (TR) (Combined Per-participant Microbiological and Clinical Success) for Gepotidacin at the Test of Cure (TOC) Visit
Description: TR at TOC (success/failure) is a measure of the overall efficacy response. A therapeutic success at TOC referred to participant who have been deemed both a microbiological success (reduction of all qualifying bacterial uropathogens recovered at BL to <10^3 colony forming units per milliliter [CFU/mL] without receiving other systemic antimicrobials [AB] before the TOC visit) and a clinical success (resolution of symptoms of acute cystitis present at BL and no new symptoms without receiving other AB before the TOC visit [or AB for uUTI on day of TOC visit]). Lack of clinical or microbiological success (including missing outcome assessments) was considered as therapeutic failure.
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S population. Participants in micro-ITT population whose baseline qualifying bacterial UP were susceptible to nitrofurantoin (NTF-S). Additionally, for the statistical analysis, therapeutic success data from the pooled global studies 204989 (NCT04020341) and 212390 (NCT04187144) were used to derive the predictive distribution, to assess the consistency of gepotidacin's therapeutic success in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin
Number analyzed (Participants) | 83
Participants
  Therapeutic Success | 69
  Therapeutic Failure | 14
Statistical Analysis 1: Comparison: Gepotidacin; As defined in Statistical Analysis Plan, consistency with the global studies is demonstrated if the success criterion for gepotidacin is set to require a therapeutic response rate greater than lower 10th percentile value of the predictive distribution; Test type: Other; Lower 10th percentile (%) = 48.2 — Lower 10th percentile of therapeutic successes was calculated from the predictive distribution

2. Secondary Outcome: Number of Participants With Therapeutic Response (TR) of Gepotidacin Compared to Nitrofurantoin at the Test of Cure (TOC) Visit - Micro-ITT NTF-S Population
Description: as for outcome 1
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S Population. Participants in the micro-ITT Population whose baseline qualifying bacterial UP were susceptible to nitrofurantoin (NTF-S).
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 83 | 25
Participants
  Therapeutic Success | 69 | 17
  Therapeutic Failure | 14 | 8

3. Secondary Outcome: Number of Participants With Clinical Outcome at the TOC Visit - Micro-ITT NTF-S Population
Description: Clinical outcome at TOC was categorized as clinical resolution, clinical improvement, clinical worsening and unable to determine. Clinical resolution at TOC was defined as resolution of signs and symptoms of acute cystitis present at BL (and no symptoms) without receiving any other AB before the TOC visit. Clinical improvement at TOC was defined as improvement (but not complete resolution) in total symptom score (CSS) from BL, without receiving any other AB before the TOC visit. Clinical worsening at TOC was defined as worsening or no change in CSS from BL or received other AB for the current infection (uUTI) before or on the date of the TOC visit. Unable to determine outcome criteria were: BL score is missing (and thus improvement/worsening cannot be determined), TOC assessment is missing, or receipt of other AB not for the current infection before the TOC visit (unless clinical worsening outcome criteria were met).
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 83 | 25
Participants
  Clinical Resolution | 71 | 19
  Clinical Improvement | 5 | 4
  Clinical Worsening | 3 | 2
  Unable To Determine | 4 | 0

4. Secondary Outcome: Number of Participants With Clinical Response at the TOC Visit - Micro-ITT NTF-S Population
Description: Clinical response at TOC was categorized as clinical success and clinical failure. Clinical success at TOC was defined as resolution of symptoms of acute cystitis present at BL (and no new symptoms), without receiving any other AB before the TOC visit. Lack of resolution, including receipt of an AB for uUTI at the TOC visit, or a missing outcome assessment was defined as Clinical Failure at TOC.
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 83 | 25
Participants
  Clinical Success | 71 | 19
  Clinical Failure | 12 | 6

5. Secondary Outcome: Number of Participants With Microbiological Outcome (MO) at the TOC Visit -Micro-ITT NTF-S Population
Description: Participant-level MO at TOC was categorized as microbiological eradication (ME), microbiological persistence (MP), microbiological recurrence (MR) and unable to determine (UTD). ME at TOC was defined as all baseline qualifying uropathogens (QUP) have an outcome of eradication at TOC (i.e., <10^3 CFU/mL without the participant receiving other systemic antimicrobials before the TOC Visit). MP at TOC was defined as at least 1 QUP has an outcome of persistence (≥10^3 CFU/mL) at TOC. MR at TOC was defined as at least 1 QUP had an outcome of recurrence and none have an outcome of persistence at TOC. UTD at TOC was defined as all QUP outcomes are UTD at TOC.
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 83 | 25
Participants
  Microbiological Eradication (ME) | 74 | 20
  Microbiological Persistence (MP) | 0 | 0
  Microbiological Recurrence (MR) | 1 | 3
  Unable To Determine (UTD) | 8 | 2

6. Secondary Outcome: Number of Participants With Microbiological Response at the TOC Visit -Micro-ITT NTF-S Population
Description: Participant-level microbiological response at TOC was categorized as microbiological success and microbiological failure. Microbiological success at TOC was defined as all baseline qualifying uropathogens (QUP) had a microbiological outcome of eradication at TOC visit. Microbiological failure was defined as lack of microbiological success, including those participants with UTD outcomes.
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 83 | 25
Participants
  Microbiological Success | 74 | 20
  Microbiological Failure | 9 | 5

7. Secondary Outcome: Number of Participants With Therapeutic Response (TR) at the TOC Visit
Description: as for outcome 1
Time Frame: At TOC visit (Days 9 to 16)
Population: Microbiological intent-to-treat multi drug resistant (Micro-ITT MDR) population included all participants in the micro-ITT Population who had any qualifying baseline bacterial uropathogens that were resistant to two or more classes of antimicrobials.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 18 | 3
Participants
  Therapeutic Success | 14 | 2
  Therapeutic Failure | 4 | 1

8. Secondary Outcome: Number of Participants With Clinical Outcome at the TOC Visit
Description: Clinical outcome at TOC was categorized as clinical resolution, clinical improvement, clinical worsening and unable to determine. Clinical resolution at TOC was defined as resolution of signs and symptoms of acute cystitis present at BL (and no symptoms) without receiving any other AB before the TOC visit. Clinical improvement at TOC was defined as improvement (but not complete resolution) in CSS from BL, without receiving any other AB before the TOC visit. Clinical worsening at TOC was defined as worsening or no change in CSS from BL or received other AB for the current infection (uUTI) before or on the date of the TOC visit. Unable to determine outcome criteria were: BL score is missing (and thus improvement/worsening cannot be determined), TOC assessment is missing, or receipt of other AB not for the current infection before the TOC visit (unless clinical worsening outcome criteria were met).
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT MDR Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 18 | 3
Participants
  Clinical Resolution | 14 | 2
  Clinical Improvement | 2 | 0
  Clinical Worsening | 1 | 1
  Unable To Determine | 1 | 0

9. Secondary Outcome: Number of Participants With Clinical Response at the TOC Visit
Description: as for outcome 4
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT MDR Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 18 | 3
Participants
  Clinical Success | 14 | 2
  Clinical Failure | 4 | 1

10. Secondary Outcome: Number of Participants With Microbiological Outcome at the TOC Visit
Description: as for outcome 5
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT MDR Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 18 | 3
Participants
  Microbiological Eradication | 16 | 2
  Microbiological Persistence | 0 | 0
  Microbiological Recurrence | 0 | 0
  Unable To Determine | 2 | 1

11. Secondary Outcome: Number of Participants With Microbiological Response at the TOC Visit
Description: as for outcome 6
Time Frame: At TOC visit (Days 9 to 16)
Population: Micro-ITT MDR Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 18 | 3
Participants
  Microbiological Success | 16 | 2
  Microbiological Failure | 2 | 1

12. Secondary Outcome: Number of Participants With Investigator Assessed Clinical Response
Description: Clinical response as assessed by investigator at TOC was categorized as clinical success and clinical failure. Clinical success at TOC was defined as sufficient resolution of acute cystitis signs and symptoms such that no additional systemic AB was required for the current infection. No apparent response to treatment, use of additional systemic AB for the current infection and death related to acute cystitis prior to the visit was considered as Clinical failure. Indeterminate/Missing was defined as participant lost to follow-up and/or the clinical assessment was not undertaken, use of confounding systemic AB for another infection, and death prior to the visit where acute cystitis was clearly noncontributory.
Time Frame: At TOC visit (Days 9 to 16)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Participants
  Clinical Success | 242 | 86
  Clinical Failure | 28 | 6
  Indeterminate/Missing | 11 | 1

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. TEAE is defined as any AE with an onset date on or after treatment start date/time. AEs were coded using Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: From first dose (Day 1) to Follow-up visit (Days 21 to 31)
Population: Safety Population included all randomized participants (except for 6 participants from the site with GCP violation) who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Participants | 201 | 18

14. Secondary Outcome: Number of Participants With Serious AEs (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Adverse events of special interest (AESI) for gepotidacin included clostridium difficile, cardiovascular & gastrointestinal events and potential acetylcholinesterase-inhibition AESIs. SAEs were coded using MedDRA.
Time Frame: From first dose (Day 1) to Follow-up visit (Days 21 to 31)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Participants
  Serious AE (SAE) | 2 | 0
  AE of Special Interest (AESIs) | 191 | 12

15. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected for urinalysis: Urine Glucose (GLU), Urine Ketones (KET), Urine Nitrite (NIT) and Urine Protein (PRO). Baseline is defined as the latest pre-dose assessment with a non-missing value. The dipstick test gives results in a semi-quantitative manner, and results can be read as Negative, Positive, 2777.55 micromole per liter (µmol/l), >=27775.5 µmol/l, 8332.65 µmol/l, 5 milligram/dl (mg/dL), 20 mg/dL, >=80 mg/dL, 300 mg/dL, 1000 mg/dL, >=5000 mg/dL indicating concentrations in the urine sample.
  In the row title (GLU, Baseline, 2777.55 micromole per liter), GLU indicates parameter, Baseline is the visit and 2777.55 micromole per liter indicates the concentration/presence in the urine sample. Data is presented in similar way for other parameters.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 280 | 93
Participants
  GLU, Baseline, 2777.55 micromole per liter | 3 | 1
  GLU, Baseline, >=27775.5 micromole per liter | 4 | 5
  GLU, Baseline, NEGATIVE | 273 | 87
  GLU, On-Therapy, 2777.55 micromole per liter: number analyzed (Participants) | 275 | 93
  GLU, On-Therapy, 2777.55 micromole per liter | 5 | 1
  GLU, On-Therapy, 8332.65 micromole per liter: number analyzed (Participants) | 275 | 93
  GLU, On-Therapy, 8332.65 micromole per liter | 2 | 0
  GLU, On-Therapy, >=27775.5 micromole per liter: number analyzed (Participants) | 275 | 93
  GLU, On-Therapy, >=27775.5 micromole per liter | 2 | 6
  GLU, On-Therapy, NEGATIVE: number analyzed (Participants) | 275 | 93
  GLU, On-Therapy, NEGATIVE | 266 | 86
  GLU, Test-of-Cure, 2777.55 micromole per liter: number analyzed (Participants) | 272 | 92
  GLU, Test-of-Cure, 2777.55 micromole per liter | 1 | 3
  GLU, Test-of-Cure, 8332.65 micromole per liter: number analyzed (Participants) | 272 | 92
  GLU, Test-of-Cure, 8332.65 micromole per liter | 1 | 0
  GLU, Test-of-Cure, >=27775.5 micromole per liter: number analyzed (Participants) | 272 | 92
  GLU, Test-of-Cure, >=27775.5 micromole per liter | 3 | 6
  GLU, Test-of-Cure, NEGATIVE: number analyzed (Participants) | 272 | 92
  GLU, Test-of-Cure, NEGATIVE | 267 | 83
  KET, Baseline, 20 milligrams per deciliter | 10 | 1
  KET, Baseline, 5 milligrams per deciliter | 26 | 13
  KET, Baseline, NEGATIVE | 244 | 79
  KET, On-Therapy, 20 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  KET, On-Therapy, 20 milligrams per deciliter | 6 | 1
  KET, On-Therapy, 5 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  KET, On-Therapy, 5 milligrams per deciliter | 22 | 7
  KET, On-Therapy, >=80 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  KET, On-Therapy, >=80 milligrams per deciliter | 0 | 1
  KET, On-Therapy, NEGATIVE: number analyzed (Participants) | 275 | 93
  KET, On-Therapy, NEGATIVE | 247 | 84
  KET, Test-of-Cure, 20 milligrams per deciliter: number analyzed (Participants) | 272 | 92
  KET, Test-of-Cure, 20 milligrams per deciliter | 1 | 0
  KET, Test-of-Cure, 5 milligrams per deciliter: number analyzed (Participants) | 272 | 92
  KET, Test-of-Cure, 5 milligrams per deciliter | 18 | 13
  KET, Test-of-Cure, NEGATIVE: number analyzed (Participants) | 272 | 92
  KET, Test-of-Cure, NEGATIVE | 253 | 79
  NIT, Baseline, NEGATIVE | 212 | 75
  NIT, Baseline, POSITIVE | 68 | 18
  NIT, On-Therapy, NEGATIVE: number analyzed (Participants) | 275 | 93
  NIT, On-Therapy, NEGATIVE | 275 | 90
  NIT, On-Therapy, POSITIVE: number analyzed (Participants) | 275 | 93
  NIT, On-Therapy, POSITIVE | 0 | 3
  NIT, Test-of-Cure, NEGATIVE: number analyzed (Participants) | 272 | 92
  NIT, Test-of-Cure, NEGATIVE | 256 | 86
  NIT, Test-of-Cure, POSITIVE: number analyzed (Participants) | 272 | 92
  NIT, Test-of-Cure, POSITIVE | 16 | 6
  PRO, Baseline, 1000 milligrams per deciliter | 43 | 19
  PRO Baseline, 300 milligrams per deciliter | 63 | 25
  PRO, Baseline, >=5000 milligrams per deciliter | 15 | 4
  PRO, Baseline, NEGATIVE | 159 | 45
  PRO, On-Therapy, 1000 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  PRO, On-Therapy, 1000 milligrams per deciliter | 12 | 1
  PRO, On-Therapy, 300 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  PRO, On-Therapy, 300 milligrams per deciliter | 46 | 17
  PRO, On-Therapy, >=5000 milligrams per deciliter: number analyzed (Participants) | 275 | 93
  PRO, On-Therapy, >=5000 milligrams per deciliter | 2 | 0
  PRO, On-Therapy, NEGATIVE: number analyzed (Participants) | 275 | 93
  PRO, On-Therapy, NEGATIVE | 215 | 75
  PRO, Test-of-Cure, 1000 milligrams per deciliter: number analyzed (Participants) | 272 | 92
  PRO, Test-of-Cure, 1000 milligrams per deciliter | 13 | 1
  PRO, Test-of-Cure, 300 milligrams per deciliter: number analyzed (Participants) | 272 | 92
  PRO, Test-of-Cure, 300 milligrams per deciliter | 24 | 11
  PRO, Test-of-Cure, >=5000 milligrams per deciliter: number analyzed (Participants) | 272 | 92
  PRO, Test-of-Cure, >=5000 milligrams per deciliter | 0 | 1
  PRO, Test-of-Cure, NEGATIVE: number analyzed (Participants) | 272 | 92
  PRO, Test-of-Cure, NEGATIVE | 235 | 79

16. Secondary Outcome: Change From Baseline (CFB) in Electrocardiograms (ECGs): Heart Rate
Description: Triplicate 12-lead ECGs (over an approximate 5 to 10 minute period) were performed using an ECG machine that automatically calculated the heart rate, measured PR, QRS, QT, and QT interval corrected for heart rate according to Fridericia's formula (QTcF). Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
beats/minute
  Baseline | 67.2 (10.18) | 70.7 (13.29)
  CFB to On-Therapy: number analyzed (Participants) | 259 | 93
  CFB to On-Therapy | -0.5 (7.84) | -3.3 (12.41)
  CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  CFB to Test-of-Cure | 0.5 (8.44) | -1.6 (12.90)

17. Secondary Outcome: Change From Baseline (CFB) in Electrocardiograms (ECGs): PR, QRS, QT and QTcF
Description: Triplicate 12-lead ECGs (over an approximate 5 to 10 minute period) were performed using an ECG machine that automatically calculated the heart rate, measured PR, QRS, QT, and QTcF. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Millisecond (msec)
  PR, Baseline | 154.9 (17.88) | 159.3 (16.68)
  PR, CFB to On-Therapy: number analyzed (Participants) | 259 | 93
  PR, CFB to On-Therapy | 1.6 (12.18) | 1.4 (9.96)
  PR, CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  PR, CFB to Test-of-Cure | 0.3 (10.47) | 0.6 (10.49)
  QRS, Baseline | 88.1 (10.06) | 89.8 (9.78)
  QRS, CFB to On-Therapy: number analyzed (Participants) | 259 | 93
  QRS, CFB to On-Therapy | 1.2 (3.77) | 0.0 (3.57)
  QRS, CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  QRS, CFB to Test-of-Cure | -0.6 (3.72) | -0.5 (3.57)
  QT, Baseline | 404.5 (28.16) | 401.1 (28.22)
  QT, CFB to On-Therapy: number analyzed (Participants) | 259 | 93
  QT, CFB to On-Therapy | 10.4 (23.67) | 4.8 (18.78)
  QT, CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  QT, CFB to Test-of-Cure | -0.7 (24.53) | 3.4 (23.23)
  QTcF, Baseline: number analyzed (Participants) | 118 | 34
  QTcF, Baseline | 418.3 (17.75) | 423.2 (17.25)
  QTcF, CFB to On-Therapy: number analyzed (Participants) | 107 | 34
  QTcF, CFB to On-Therapy | 10.3 (13.44) | 1.8 (10.82)
  QTcF, CFB to Test-of-Cure: number analyzed (Participants) | 113 | 34
  QTcF, CFB to Test-of-Cure | 1.3 (12.09) | 3.6 (11.66)

18. Secondary Outcome: Change From Baseline (CFB) in Vital Sign: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Millimeters of mercury (mmHg)
  Diastolic Blood Pressure, Baseline | 72.8 (11.98) | 74.5 (12.60)
  Diastolic Blood Pressure, CFB to On-Therapy: number analyzed (Participants) | 274 | 93
  Diastolic Blood Pressure, CFB to On-Therapy | -2.6 (9.45) | -2.1 (9.36)
  Diastolic Blood Pressure, CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  Diastolic Blood Pressure, CFB to Test-of-Cure | -2.4 (9.76) | -3.9 (9.64)
  Systolic Blood Pressure, Baseline | 118.2 (18.10) | 118.7 (18.38)
  Systolic Blood Pressure, CFB to On-Therapy: number analyzed (Participants) | 274 | 93
  Systolic Blood Pressure, CFB to On-Therapy | -3.1 (12.20) | -3.3 (13.32)
  Systolic Blood Pressure, CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  Systolic Blood Pressure, CFB to Test-of-Cure | -3.7 (11.63) | -4.1 (11.35)

19. Secondary Outcome: Change From Baseline (CFB) in Vital Sign: Temperature
Description: Temperature was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Celsius
  Baseline | 36.49 (0.367) | 36.44 (0.365)
  CFB to On-Therapy: number analyzed (Participants) | 274 | 93
  CFB to On-Therapy | -0.05 (0.453) | -0.03 (0.425)
  CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  CFB to Test-of-Cure | -0.07 (0.397) | -0.02 (0.396)

20. Secondary Outcome: Change From Baseline (CFB) in Vital Sign: Pulse Rate
Description: Pulse rate was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
beats/minute
  Baseline | 69.7 (10.79) | 72.2 (10.65)
  CFB to On-Therapy: number analyzed (Participants) | 274 | 93
  CFB to On-Therapy | 2.4 (10.36) | 1.4 (10.66)
  CFB to Test-of-Cure: number analyzed (Participants) | 272 | 92
  CFB to Test-of-Cure | 0.4 (9.30) | -0.5 (11.54)

21. Secondary Outcome: Plasma Concentrations of Gepotidacin
Description: Blood samples were collected for plasma concentration of Gepotidacin.
Time Frame: Baseline (Day 1 at 0-2h & >2h Post dose), Day 2 to 5 at Pre-dose, 0-2h & >2h Post Dose
Population: Pharmacokinetic (PK) Population included all randomized participants (excluding 6 participants from a site with GCP violation), who received at least 1 dose of Gepotidacin and had at least 1 non-missing plasma concentration (Non-quantifiable values were considered as non-missing). Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram/ milliliter (ng/mL)
Arm/Group | Gepotidacin
Number analyzed (Participants) | 267
Nanogram/ milliliter (ng/mL)
  Baseline, POST-DOSE, Day 1, 0-2h | 5210.23 (3428.432)
  Baseline, POST-DOSE, Day 1, >2h: number analyzed (Participants) | 13
  Baseline, POST-DOSE, Day 1, >2h | 5251.54 (2097.649)
  On-Therapy, PRE-DOSE, Day 2-5, pre-dose: number analyzed (Participants) | 247
  On-Therapy, PRE-DOSE, Day 2-5, pre-dose | 1960.14 (16752.767)
  On-Therapy, POST-DOSE, Day 2-5, 0-2h: number analyzed (Participants) | 245
  On-Therapy, POST-DOSE, Day 2-5, 0-2h | 17548.67 (124724.240)
  On-Therapy, POST-DOSE, Day 2-5, >2h: number analyzed (Participants) | 5
  On-Therapy, POST-DOSE, Day 2-5, >2h | 5976.40 (5142.635)

22. Secondary Outcome: Urine Concentrations of Gepotidacin
Description: Urine samples were collected for urine concentration of Gepotidacin.
Time Frame: Baseline (Day 1 at 0-2h & >2h Post dose), Day 2 to 5 at Pre-dose, 0-2h & >2h Post Dose
Population: Pharmacokinetic (PK) Population included all randomized participants (excluding 6 participants from a site with GCP violation), who received at least 1 dose of Gepotidacin and had at least 1 non-missing urine concentration (Non-quantifiable values were considered as non-missing). Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Microgram/ milliliter (ug/mL)
Arm/Group | Gepotidacin
Number analyzed (Participants) | 250
Microgram/ milliliter (ug/mL)
  Baseline, POST-DOSE, Day 1, 0-2h | 506.988 (914.3140)
  Baseline, POST-DOSE, Day 1, >2h: number analyzed (Participants) | 28
  Baseline, POST-DOSE, Day 1, >2h | 600.729 (644.2265)
  On-Therapy, PRE-DOSE, Day 2-5, pre-dose: number analyzed (Participants) | 248
  On-Therapy, PRE-DOSE, Day 2-5, pre-dose | 492.096 (565.8822)
  On-Therapy, POST-DOSE, Day 2-5, 0-2h: number analyzed (Participants) | 231
  On-Therapy, POST-DOSE, Day 2-5, 0-2h | 901.554 (1451.8781)
  On-Therapy, POST-DOSE, Day 2-5, >2h: number analyzed (Participants) | 19
  On-Therapy, POST-DOSE, Day 2-5, >2h | 1138.900 (1429.7998)

23. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameters - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, and Platelets at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, and platelets. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per Liter (10^9 cells/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 245 | 84
Giga cells per Liter (10^9 cells/L)
  Basophils, Baseline: number analyzed (Participants) | 243 | 84
  Basophils, Baseline | 0.050 (0.0238) | 0.051 (0.0223)
  Basophils, CFB to On-Therapy: number analyzed (Participants) | 231 | 78
  Basophils, CFB to On-Therapy | -0.004 (0.0194) | -0.001 (0.0152)
  Basophils, CFB to Test-of-Cure: number analyzed (Participants) | 220 | 81
  Basophils, CFB to Test-of-Cure | -0.001 (0.0192) | -0.002 (0.0135)
  Eosinophils, Baseline: number analyzed (Participants) | 243 | 84
  Eosinophils, Baseline | 0.134 (0.1199) | 0.121 (0.0977)
  Eosinophils, CFB to On-Therapy: number analyzed (Participants) | 231 | 78
  Eosinophils, CFB to On-Therapy | 0.008 (0.0567) | 0.011 (0.0500)
  Eosinophils, CFB to Test-of-Cure: number analyzed (Participants) | 220 | 81
  Eosinophils, CFB to Test-of-Cure | 0.028 (0.0862) | 0.023 (0.0630)
  Lymphocytes, Baseline: number analyzed (Participants) | 243 | 84
  Lymphocytes, Baseline | 1.657 (0.5001) | 1.727 (0.5203)
  Lymphocytes, CFB to On-Therapy: number analyzed (Participants) | 231 | 78
  Lymphocytes, CFB to On-Therapy | -0.044 (0.3958) | 0.075 (0.4024)
  Lymphocytes, CFB to Test-of-Cure: number analyzed (Participants) | 220 | 81
  Lymphocytes, CFB to Test-of-Cure | -0.054 (0.4698) | 0.111 (0.4414)
  Monocytes, Baseline: number analyzed (Participants) | 243 | 84
  Monocytes, Baseline | 0.388 (0.1474) | 0.375 (0.1394)
  Monocytes, CFB to On-Therapy: number analyzed (Participants) | 231 | 78
  Monocytes, CFB to On-Therapy | -0.057 (0.1457) | -0.059 (0.1584)
  Monocytes, CFB to Test-of-Cure: number analyzed (Participants) | 220 | 81
  Monocytes, CFB to Test-of-Cure | -0.049 (0.1503) | -0.033 (0.1393)
  Neutrophils, Baseline: number analyzed (Participants) | 242 | 84
  Neutrophils, Baseline | 4.805 (2.1102) | 4.684 (2.0992)
  Neutrophils, CFB to On-Therapy: number analyzed (Participants) | 231 | 78
  Neutrophils, CFB to On-Therapy | -1.530 (1.8841) | -1.477 (1.9168)
  Neutrophils, CFB to Test-of-Cure: number analyzed (Participants) | 219 | 81
  Neutrophils, CFB to Test-of-Cure | -1.713 (2.2275) | -1.493 (2.1633)
  Platelets, Baseline: number analyzed (Participants) | 245 | 83
  Platelets, Baseline | 261.0 (58.37) | 253.6 (56.80)
  Platelets, CFB to On-Therapy: number analyzed (Participants) | 232 | 76
  Platelets, CFB to On-Therapy | 5.7 (25.42) | 2.6 (21.53)
  Platelets, CFB to Test-of-Cure: number analyzed (Participants) | 224 | 79
  Platelets, CFB to Test-of-Cure | 3.3 (34.80) | 4.2 (37.13)

24. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter-Hemoglobin Level at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of hemoglobin level. Baseline is defined as the latest pre-dose assessment with a non-missing value
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 246 | 85
Grams per Liter (g/L)
  Baseline | 128.6 (10.70) | 128.0 (10.91)
  CFB to On-Therapy: number analyzed (Participants) | 235 | 79
  CFB to On-Therapy | -1.3 (6.01) | -1.0 (5.61)
  CFB to Test-of-Cure: number analyzed (Participants) | 226 | 82
  CFB to Test-of-Cure | -2.3 (6.22) | -2.9 (6.39)

25. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter- Hematocrit Level at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of hematocrit level. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 246 | 85
Proportion of red blood cells in blood
  Baseline | 0.4355 (0.04242) | 0.4308 (0.05058)
  CFB to On-Therapy: number analyzed (Participants) | 235 | 79
  CFB to On-Therapy | -0.0047 (0.03252) | 0.0067 (0.03567)
  CFB to Test-of-Cure: number analyzed (Participants) | 226 | 82
  CFB to Test-of-Cure | -0.0082 (0.03441) | -0.0038 (0.03533)

26. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter- Erythrocytes Count at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of erythrocytes count. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Tera cells per Liter (10^12 cells/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 246 | 85
Tera cells per Liter (10^12 cells/L)
  Baseline | 4.302 (0.3650) | 4.245 (0.3758)
  CFB to On-Therapy: number analyzed (Participants) | 235 | 79
  CFB to On-Therapy | -0.040 (0.2021) | -0.025 (0.1887)
  CFB to Test-of-Cure: number analyzed (Participants) | 226 | 82
  CFB to Test-of-Cure | -0.085 (0.2157) | -0.098 (0.2218)

27. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter - Mean Corpuscular Hemoglobin (MCH) at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of MCH. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 246 | 85
Picogram (pg)
  Baseline | 29.97 (2.062) | 30.26 (2.170)
  CFB to On-Therapy: number analyzed (Participants) | 235 | 79
  CFB to On-Therapy | -0.03 (0.536) | -0.05 (0.519)
  CFB to Test-of-Cure: number analyzed (Participants) | 226 | 82
  CFB to Test-of-Cure | 0.04 (0.613) | 0.00 (0.629)

28. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter - Mean Corpuscular Volume (MCV) at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of MCV. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 246 | 85
Femtoliter (fL)
  Baseline | 101.48 (8.607) | 101.65 (10.185)
  CFB to On-Therapy: number analyzed (Participants) | 235 | 79
  CFB to On-Therapy | -0.16 (6.300) | 2.40 (7.634)
  CFB to Test-of-Cure: number analyzed (Participants) | 226 | 82
  CFB to Test-of-Cure | 0.08 (6.740) | 1.61 (7.071)

29. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Calcium, Glucose, Potassium, Magnesium, Phosphate, Sodium, and Urea Nitrogen Levels at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of clinical chemistry parameters. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
millimoles per liter (mmol/L)
  Calcium, Baseline | 2.319018 (0.0816980) | 2.314716 (0.0868299)
  Calcium, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Calcium, CFB to On-Therapy | -0.004536 (0.0766926) | -0.012341 (0.0695672)
  Calcium, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Calcium, CFB to Test-of-Cure | -0.032315 (0.0855497) | -0.029885 (0.0860459)
  Glucose, Baseline | 5.196605 (1.1351979) | 5.458483 (1.7589320)
  Glucose, CFB to On-Therapy: number analyzed (Participants) | 274 | 93
  Glucose, CFB to On-Therapy | 0.248377 (1.3575780) | 0.423189 (1.3092369)
  Glucose, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Glucose, CFB to Test-of-Cure | 0.057763 (1.1507851) | 0.156160 (1.2016889)
  Potassium, Baseline: number analyzed (Participants) | 280 | 92
  Potassium, Baseline | 4.13 (0.339) | 4.16 (0.364)
  Potassium, CFB to On-Therapy: number analyzed (Participants) | 273 | 91
  Potassium, CFB to On-Therapy | 0.05 (0.329) | 0.02 (0.310)
  Potassium, CFB to Test-of-Cure: number analyzed (Participants) | 269 | 90
  Potassium, CFB to Test-of-Cure | 0.00 (0.365) | 0.04 (0.370)
  Magnesium, Baseline | 0.862 (0.0605) | 0.860 (0.0632)
  Magnesium, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Magnesium, CFB to On-Therapy | -0.004 (0.0555) | -0.010 (0.0519)
  Magnesium, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Magnesium, CFB to Test-of-Cure | -0.010 (0.0569) | -0.014 (0.0651)
  Phosphate, Baseline | 1.184963 (0.1593757) | 1.206882 (0.1775576)
  Phosphate, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Phosphate, CFB to On-Therapy | 0.009746 (0.1600765) | -0.031943 (0.1706300)
  Phosphate, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Phosphate, CFB to Test-of-Cure | 0.019541 (0.1736731) | 0.036903 (0.1985578)
  Sodium, Baseline | 139.8 (2.25) | 139.8 (2.13)
  Sodium, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Sodium, CFB to On-Therapy | 0.1 (2.33) | -0.2 (2.38)
  Sodium, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Sodium, CFB to Test-of-Cure | 0.1 (2.52) | 0.2 (2.42)
  Urea Nitrogen, Baseline | 4.3094 (1.32217) | 4.4145 (1.33139)
  Urea Nitrogen, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Urea Nitrogen, CFB to On-Therapy | -0.0948 (0.98541) | -0.1689 (0.85458)
  Urea Nitrogen, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Urea Nitrogen, CFB to Test-of-Cure | 0.1423 (1.07780) | 0.1177 (0.91259)

30. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Serum Chloride at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliequivalents per liter (mEq/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Milliequivalents per liter (mEq/L)
  Baseline | 102.3 (2.21) | 102.4 (2.38)
  CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  CFB to On-Therapy | 0.8 (2.23) | 0.3 (2.36)
  CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  CFB to Test-of-Cure | 1.0 (2.46) | 0.6 (2.58)

31. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Direct Bilirubin, Total Bilirubin and Creatinine Levels at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per Liter (umol/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
micromoles per Liter (umol/L)
  Direct Bilirubin, Baseline | 3.4498 (0.23845) | 3.4329 (0.10767)
  Direct Bilirubin, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Direct Bilirubin, CFB to On-Therapy | -0.0056 (0.24374) | -0.0129 (0.10767)
  Direct Bilirubin, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Direct Bilirubin, CFB to Test-of-Cure | -0.0063 (0.20804) | -0.0113 (0.11053)
  Total Bilirubin, Baseline | 7.0731 (4.66102) | 6.0420 (3.11713)
  Total Bilirubin, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Total Bilirubin, CFB to On-Therapy | -0.4079 (4.14317) | 0.3163 (3.23527)
  Total Bilirubin, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Total Bilirubin, CFB to Test-of-Cure | -0.1723 (4.23182) | 0.2988 (2.99514)
  Creatinine, Baseline | 50.964 (8.7527) | 52.280 (11.9212)
  Creatinine, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Creatinine, CFB to On-Therapy | 3.632 (6.6395) | -1.426 (6.9325)
  Creatinine, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Creatinine, CFB to Test-of-Cure | 0.620 (7.9007) | 0.000 (7.0965)

32. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Creatinine Clearance at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter/second (mL/s)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Milliliter/second (mL/s)
  Baseline | 1.8346749 (0.58199842) | 1.8690338 (0.63944090)
  CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  CFB to On-Therapy | -0.1155781 (0.27838072) | 0.0331548 (0.28390850)
  CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  CFB to Test-of-Cure | -0.0284139 (0.27653678) | -0.0111724 (0.24923906)

33. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Albumin and Protein Levels at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
gram per Liter (g/L)
  Albumin, Baseline | 44.7 (2.51) | 44.1 (2.91)
  Albumin, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Albumin, CFB to On-Therapy | -0.4 (2.19) | -0.3 (2.11)
  Albumin, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Albumin, CFB to Test-of-Cure | -1.3 (2.36) | -1.2 (2.26)
  Protein, Baseline | 70.6 (4.18) | 70.7 (4.46)
  Protein, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  Protein, CFB to On-Therapy | -0.8 (3.50) | -0.7 (3.71)
  Protein, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  Protein, CFB to Test-of-Cure | -2.1 (3.80) | -2.3 (3.72)

34. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters - Alkaline Phosphatase (ALP) and Alanine Aminotransferase (ALT) Levels at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
International Units per Liter (IU/L)
  ALP, Baseline | 68.9 (22.09) | 68.4 (22.18)
  ALP, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  ALP, CFB to On-Therapy | -0.1 (6.10) | -0.4 (8.10)
  ALP, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  ALP, CFB to Test-of-Cure | -2.9 (7.12) | -3.1 (9.28)
  ALT, Baseline | 17.0 (16.80) | 16.7 (11.11)
  ALT, CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  ALT, CFB to On-Therapy | 1.2 (6.16) | -0.2 (3.28)
  ALT, CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  ALT, CFB to Test-of-Cure | 0.6 (12.59) | -1.1 (5.98)

35. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameter - Aspartate Aminotransferase (AST) Levels at On Therapy and Test of Cure Visit
Description: as for outcome 29
Time Frame: Baseline (Day 1), On-Therapy (Days 2 to 5), and at TOC visit (Days 9 to 16)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 281 | 93
Units per Liter (U/L)
  Baseline | 20.1 (17.26) | 18.7 (7.12)
  CFB to On-Therapy: number analyzed (Participants) | 275 | 93
  CFB to On-Therapy | 0.4 (11.28) | 0.0 (3.85)
  CFB to Test-of-Cure: number analyzed (Participants) | 271 | 91
  CFB to Test-of-Cure | 0.8 (16.01) | -0.2 (4.49)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from first dose (Day 1) to follow-up visit (Days 21 to 31).
Description: Safety Population
Arm/Group | Gepotidacin | Nitrofurantoin
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/93
Serious Adverse Events (participants affected / at risk) | 2/281 | 0/93
Other Adverse Events (participants affected / at risk) | 174/281 | 8/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=281) | Nitrofurantoin (N=93)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=281) | Nitrofurantoin (N=93)
Diarrhoea (Gastrointestinal disorders) | 167 (175) | 7 (9)
Nausea (Gastrointestinal disorders) | 35 (35) | 2 (2)

LIMITATIONS AND CAVEATS:
GlaxoSmithKline (GSK) was informed of suspected GCP violations in a Japanese site management organization which provided site management services to one of the sites for this study, at which 6 participants were enrolled (5 gepotidacin participants; 1 nitrofurantoin participant). These 6 participants were excluded from the analysis due to data integrity issues including undeniable suspected data falsification that resulted in unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT05630833/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT05630833/SAP_001.pdf